CLINICAL TRIAL: NCT04715789
Title: EFFECT OF COGNITIVE BEHAVIOURALTHERAPY IN TREATMENT OF CHRONIC NON-SPECIFIC LOW BACK PAIN
Brief Title: COGNITIVE BEHAVIOURAL THERAPY FOR TREATMENT OF CHRONIC NON-SPECIFIC LOW BACK PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohmed yehia elabd hasan, phyisical therapist at qena oncology center, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COGNITIVE BEHAVIOURAL THERAPY
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain
Keywords: graded eposure and activity
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Clinical trial controled study with double blind procedures for (main investigator) for treatment interventions and (research assistance) for assessment interventions.
Who Masked: Care Provider, Investigator
Masking Description: The main investigator will perform the physical therapy program after referral by Blind assessor after assessment.
  Main investigator start the treatment based on the randomization made by the software after the referral so he will not know the assessment results before and after he treatment and the assessor will not know the randomization results and the patient group selected for treatment
  So this procedures will be done by double blind procedure for the main investigator and research assistance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy intervention (Experimental): 1. core stability exercises:
     1. Multifidus exercises
     2. Frontal & Side Plank exercise
     3. Pelvic floor exercises
     4. abdominal exercises
  2. Strengthening exercises
     1. Bridging
     2. straight leg raise
     3. gluteus medius strength
     4. gluteus maximus strengthening for about 20 min to 30 min to strength back and proximal hip control muscles
  Interventions: Behavioral: graded exposure and activity
- graded exposure and graded activity in addition to phycal therapy intervention (Experimental): 1. Graded exposure:This approach followed a model where the patient was gradually exposed to previously pain provocative, feared and or avoided tasks. These activities are started at a diminished level that elicits minimal amounts of fear and then gradually increased to situations that elicit larger amounts of fear patients are asked to create a hierarchy of feared activities. The exposure starts with the least feared activity, and the therapist helps the patient appraise the exposure and its consequences and then address irrational and counterproductive beliefs, leading to reductions in the anxiety associated with the activity
  2. Graded activity exercises: The new postural and movement behaviors were integrated into each person's nominated pain provocative functional activities linked to their goals in order to generalize learning and build self-efficacy the program focuses on functional activities for about 10 min before physical therapy program (strengthening)
  Interventions: Behavioral: graded exposure and activity

INTERVENTIONS:
Behavioral: graded exposure and activity — 1. Graded exposure: This approach followed a model where the patient was gradually exposed to previously pain provocative, feared and or avoided tasks. These activities are started at a diminished level that elicits minimal amounts of fear and then gradually increased to situations that elicit larger amounts of fear patients are asked to create a hierarchy of feared activities. The exposure starts with the least feared activity, and the therapist helps the patient appraise the exposure and its consequences and then address irrational and counterproductive beliefs, leading to reductions in the anxiety associated with the activity
  2. Graded activity exercises: The new postural and movement behaviors were integrated into each person's nominated pain provocative functional activities linked to their goals in order to generalize learning and build self-efficacy the program focuses on functional activities and progresses in a time contingent manner

SUMMARY:
To explore the effect of adding cognitive-behavioral therapy to physical therapy interventions in patients with chronic non-specific back pain.

DETAILED DESCRIPTION:
Studies suggest that patients with LBP benefited when standard rehabilitation approaches were supplemented with graded exercise . There is adequate information to allow clinical implementation of graded exercise by physical therapists, In contrast, there is less information available for physical therapy implementation of graded exposure. LBP rehabilitation based on graded exposure principles Therefore, the purpose of this study is to review the available evidence for graded exposure and to describe physical therapy application of graded exposure for patients enrolled in clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age between 25-40 years.
2. Patients have persistent Chronic Non-specific LBP for at least 3 months with or without leg pain. Leg pain won't exceeds mechanical behaviors.
3. Score of 24 fear avoidance questionnaire.
4. Symptoms of hypersensitivity, secondary punctate or pressure hyperalgesia and fear of movement as a central sensitization symptoms

Exclusion Criteria:

* 1-History of previous back surgery. 2- History of previous hip, knee or ankle surgeries. 3- Systemic inflammatory diseases. 4-Tumors. 5-Red flags of back pain 6-Patients with disc pathology and radicular pain 7- spinal fracture or spinal surgery 8- systemic disease or TB of spine widespread constant non-specific pain disorder, pain without a clear mechanical behavior

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Arabic ODI for function | 5 minutes
  a)ODI ASSESMENT: Patient-completed questionnaire which gives a percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain. In pre session and after end of sessions This Questionnaire examines perceived level of disability in 10 everyday activities of daily living.
  The 6 statements are scored from 0 to 5 with the first statement scoring 0 through to the last at5 If all 10 sections are completed the score is calculated as follows: if 16 (total scored) out of 50 (total possible score) x 100 = 32% Scores: 1- (0% to 20%): minimal disability 2-(21%-40%: moderate disability) 3- (41%-60%): severe disability 4-(61%-80%: crippled) 5-(81%-100%) These patients are either bed-bound or exaggerating their symptoms

SECONDARY OUTCOMES:
Numerical rating scale | 5 minutes
  patient will sign the degree of pain from(0to 10) the assessment will be done in pretreatment and post treatment as an outcome measure for pain intensity.
Tape measurement | 5 minutes
  the patient will be informed about the rules of upright position and asked to position himself in front of the mirror. This posture was recorded as the upright position of the patient and the measurements for the posture analysis were recorded by means of a tape measure from c7 to s2
Fear avoidance belief questionnaire | 5 minutes
  The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. the patient fill the questionnaire in first session and at last session

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: https://pubmed.ncbi.nlm.nih.gov/ — https://pubmed.ncbi.nlm.nih.gov/